CLINICAL TRIAL: NCT05590598
Title: Prospective, Multicenter, Open-label, Randomized, Parallel, Clinical Study for Assessment of Comparative Efficacy and Safety of Azelastine +Mometasone , Nasal Spray, 140 mcg + 50 mcg, (Sandoz d.d., Slovenia) and Momat Rino Advance, Nasal Spray, 140 mcg + 50 mcg, (Glenmark, India) Administered as a Monotherapy to Patients With Seasonal Allergic Rhinitis.
Brief Title: Efficacy and Safety of Azelastine +Mometasone , Nasal Spray, 140 mcg + 50 mcg, (Sandoz d.d., Slovenia) and Momat Rino Advance, Nasal Spray, 140 mcg + 50 mcg, (Glenmark, India) Administered as a Monotherapy to Patients With Seasonal Allergic Rhinitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAN-0727
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Azelastine + Mometasone, nasal spray (Experimental): Participants will receive test product Azelastine + Mometasone, nasal spray, 140 mcg + 50 mcg/dose (Sandoz d.d., Slovenia), one actuation in each nostril twice daily, morning and evening (recommended interval between administrations is approximately 12 hours), for 14 consecutive days.
  Interventions: Combination Product: Azelastine + Mometazone, nasal spray
- Group 2: Momat Rhino Advance, nasal dosed spray (Active Comparator): Participants will receive reference product Momat Rhino Advance, nasal dosed spray, 140 mcg + 50 mcg mcg/dose (Glenmark Pharmaceuticals Limited., India), one actuation in each nostril twice daily, morning and evening (recommended interval between administrations is approximately 12 hours), for 14 consecutive days.
  Interventions: Combination Product: Momat Rhino Advance

INTERVENTIONS:
Combination Product: Azelastine + Mometazone, nasal spray — 140 mcg + 50 mcg/dose (Sandoz d.d., Slovenia), one actuation in each nostril twice daily, morning and evening (recommended interval between administrations is approximately 12 hours), for 14 consecutive days.
  Arms: Group 1: Azelastine + Mometasone, nasal spray
Combination Product: Momat Rhino Advance — 140 µg + 50 µg/dose - one actuation into each nostril twice daily - morning and evening (interval between administrations is 12 hrs), corresponding to 560 µg/day of azelastine and 200 µg/day of mometasone for 14 consecutive days
  Arms: Group 2: Momat Rhino Advance, nasal dosed spray

SUMMARY:
Prospective, multicenter, open, randomized, parallel, clinical study for assessment of comparative efficacy and safety of Azelastine +Mometasone Sandoz (main group) and Momat Rino Advance (control group) administered as a monotherapy to patients with seasonal allergic rhinitis (SAR).

DETAILED DESCRIPTION:
The maximum observation period will be 22 days. Study periods

* Screening (Visit 1): 1 day prior to Run-In period start (-4 day before study treatment ).
* Run-In Period: 3 days prior to first administration of test product/reference product (-3 to -1 days before study treatment).
* Randomization (Visit 2): assignment of test product/reference product to the patient (study treatment: day 1).
* Administration of test product/reference product within Study days 1 to 14 and observation at Visits 2, 3, 4 which correspond to study days 1, 7, 15, respectively.
* Period of follow-up (Visit 5): 36-96 h after last administration of test product/reference product. Performed in a form of a phone call (study treatment: days 16-18).

Patients meeting the inclusion criteria and not meeting the non-inclusion criteria will be randomized into 2 groups in a 1:1 ratio.

Dose of test product/reference product and dosing regimen used in this study are based on PIL of original product Momat Rino Advance approved by Ministry of Healthcare of the Russian Federation which is used in this study as a reference product.

Test product and reference product in this study will be administered according to the following regimen:

Group 1 (n=236) will receive test product Azelastine + Mometasone, nasal spray, 140 mcg + 50 mcg/dose (Sandoz d.d., Slovenia), one actuation in each nostril twice daily, morning and evening (recommended interval between administrations is approximately 12 hours), for 14 consecutive days.

Group 2 (n=236) will receive reference product Momat Rhino Advance, nasal dosed spray, 140 mcg + 50 mcg mcg/dose (Glenmark Pharmaceuticals Limited., India), one actuation in each nostril twice daily, morning and evening (recommended interval between administrations is approximately 12 hours), for 14 consecutive days

All study procedures for both groups at each phase of study are identical.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following criteria will be included in the study and allocated to treatment groups:

* 18 to 65 years old inclusive, male and female;
* voluntarily signed informed consent for participation in this clinical study;
* presence of confirmed moderate or severe seasonal allergic rhinitis occurring during pollen/allergen season of at least 24 months prior to enrollment in the study;
* presence of nasal symptoms of SAR (nasal congestion, rhinorrhea, nasal itching, sneezing): total score as per scale of reflective Total Nasal Symptoms Score (r-TNSS) at least 6: wherein, nasal congestion - at least 2 scores, as well as at least 2 scores in assessment of at least one of other three symptoms at Screening Visit and Visit 2;
* presence of documented positive result for dermic allergy test and/or serology allergen-specific IgE test performed for one or more allergens 12 months or earlier prior to enrollment to this study (patients should have positive skin tests and/or serology allergen-specific IgE test at least with one allergen, specific to the season during which clinical trial is conducted);
* fertile females shall have negative pregnancy test at screening (except for the women after surgical sterilization or with 2 year and more period of menopause);
* for women of child-bearing potential - consent to use one of following methods of effective contraception for the duration of study, as well for 30 days after the study end: Total abstinence. Oral contraceptives (combination medications containing progestagen or only progestagen).

Injection progestogen. Implants with levonorgestrel. Estrogen containing vaginal ring. Skin patch with contraceptive. Intrauterine device (IUD) or intrauterine system (IUS) that complies with efficacy criteria as stated in PIL.

* Male partner is sterile (vasectomy with documented azoospermia) prior to female enrollment into the study based on condition that this partner is the only partner for this patient. For this definition "documented" is related to the result of medical examination by Investigator/Patient's Responsible Party or medical history review for assessment of enrollment to the study received orally by the patient or from medical record of the patient.
* Double barrier method: condom or occlusive cap (diaphragm or cervical/camerated cap) plus spermicide (foam/gel/film/cream/suppository);
* for male subjects: consent to follow with the female partner adequate contraception method for the duration of participation in the study from beginning to the end, as well as for 30 days after the end of the study;
* absence of somatic diseases of unstable severe character or in the phase of decompensation;
* ability to understand information about clinical study, readiness to follow requirements of study protocol, ability to use dosed nasal spray individually and assess symptoms of seasonal allergic rhinitis with the help of rating scale.

Non-inclusion Criteria:

Patients related to any of the following groups will not be included in the study:

* Patients with hypersensitivity to mometasone/ azelastine and/or excipients containing in test product/reference product.
* Patients with anaphylaxis and/or other severe local reaction(s) to skin test documented in medical history (scarification tests/prick tests).
* Negative or controversial result of dermic allergy tests and/or serology allergen-specific IgE test.
* Patients with asthma in medical history with regard to which during last 2 years regular therapy was required; patients with light asthma connected with physical exercises are enrolled to the study based on condition that it is treated only with beta-adrenergic agonists of short action.
* Patients with nasal cavity and/or paranasal sinuses diseases, including:

acute or chronic sinusitis; non-allergic rhinitis, fungal and bacterial infection, as well as with purulent discharge from nose for 30 days, virus infections for 7 days prior to administration of compared products; perennial allergic rhinitis; rhinitis medicamentosa; atrophic rhinitis; nasal polyps with breathing difficulty; erosion and ulcer of nasal mucosa; significant deflection of nasal septum, other structural changes in nasal cavity that preclude from correct air transit; nasal bleeding tendency.

* Patients who resumed immune therapy (including locally administered products); or patients who had changes in the schedule of allergen-specific immune therapy in the period of 30 days prior to Screening visit or patients who have planned to start immune therapy during participation in the study.
* Patients who had surgery of nasal cavity or paranasal sinuses, nasal trauma, ocular surgery or eye trauma less than 12 months (1 year) prior to Screening visit
* Treatment of oral cavity candidiasis 30 days prior to Screening visit or patients with oral cavity candidiasis at the moment of Screening visit.
* Patients with past or unstable concomitant diseases or clinical states that preclude patient from enrollment to the study (decision is taken by investigator), including:

respiratory diseases (for example, pulmonary tuberculosis, severe asthma, airway hyperreactivity, other broncho-obstructive diseases); untreated fungal, bacterial, virus infections (including herpes simplex); dysfunction of hypothalamo-pituitary-adrenal axis; diabetes; arterial hypertension; oncology diseases; mental illnesses, administration of monoaminooxidase inhibitors (IMAO), tricyclic antidepressants; angle-closure glaucoma, increased intraocular pressure, posterior subcapsular cataract; eye Herpes simplex or other eye infections in the period of 14 days prior to Screening visit; Hepatitis B or C, syphilis; HIV infected patients;

* Varicella or rubeola or contacts with patients diagnosed with varicella or rubeola in the period of 30 days prior to Screening visit.
* Administration of any glucocorticosteroid ophthalmologic products in the period of 14 days or nasally inhaled, systematic glucocorticosteroids in the period of 30 days prior to Screening visit. Hormonal contraception or hormonal replacement therapy is acceptable in case that patient has stable dosing regimen for at least 30 days prior to Screening visit or has stable dosing regimen for the period of the study.
* Administration of nasal or other systemic first generation antihistamines, antileukotrienes or other decongestants in the period of 3 days prior to Screening visit.
* Administration of nasal or systemiс second generation antihistamines in the period of 10 days prior to Screening visit.
* Administration of medicinal products containing cromoglicic acid in the period of 14 days prior to Screening visit.
* Administration of any tricyclic antidepressants in the period of 30 days prior to Screening visit.
* Patients with attention deficit disorder without stable therapy regime in the period of 30 days prior to Screening visit or planning to change therapy regime in the period of study.
* ASIT (allergen-specific immunotherapy) by seasonal allergen which was the cause of allergic rhinitis for the patient in the period of 6 months prior to Screening visit.
* Seasonal allergic rhinitis or perennial allergic rhinitis not responding to glucocorticosteroids documented in medical history;
* Patients that are not willing to refrain from any systemic or local (i.ae. nasal, ophthalmologic) vasoconstrictive, decongestant products and/or other products for treatment of SAR from the moment of informed consent signed and prior to Follow-up visit;
* Patients with history or presence of drug/alcohol abuse.
* Pregnant or breast-feeding females.
* Male patients and female patients with reproductive potential that refuse to use adequate contraception methods during the study and for 30 days after last administration of compared products.
* Patients who had surgery in the period of 30 days prior to Screening visit and patients that will have surgeries during the study (prior to the end of Follow-up visit), as well as diagnostic procedures or visiting in-patient clinic.
* Patients participating in other clinical studies of medicinal products at the moment of Screening visit or that participated in them in the period of 30 days prior to Screening visit.
* Possibility of traveling outside the region of permanent residence during the study conduct.
* Any diseases or circumstances which, in Investigator's opinion, can prevent subject from participation in the study or which can present danger to the subject's participation in the study.
* Positive tests for markers of viral hepatitis B, C, syphilis, HIV infection, PCR test for coronavirus SARS-CoV-2.
* Positive breath alcohol vapor test.
* Positive urine test for narcotic drugs and psychotropic substances (cocaine, cannabis, amphetamine, barbiturates, benzodiazepines and opioids).

Exclusion Criteria:

The subject's participation will be terminated if any of the following causes occurs:

* The occurrence of any disease or condition during the study that worsens the patient's prognosis and makes it impossible for the patient to participate further in the clinical trial.
* The need to prescribe prohibited concomitant therapy.
* A positive PCR test for SARS-CoV-2.
* Pregnancy of the patient.
* Violation of the Study Protocol: Erroneous inclusion of a patient who does not meet the inclusion criteria and/or meets the non-inclusion criteria; taking forbidden therapy; Other violations of the Protocol, which in the opinion of the Investigator are significant.
* Patient's refusal to participate in the study.
* Other administrative reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Mean total score change as per scale r-TNSS (AM/PM) with initial total score | Day 1, 7 and 15 post treatment
  r-TNSS (reflective Total Nasal Symptom Score) consists of 4 symptom scores (Nasal congestion, Runny nose, Itchy nose, Sneezing), each of which can be scored on a 4-point scale (0-3). Higher scores mean a more severe symptom.
  By its nature, the total index r-TNSS is a rank indicator, it is an integer from the range from 0 to 12 points. As a working indicator, the average between the morning and evening values is used.
  As a measure of the effect of the drug, the change in the index relative to the initial value is used. Baseline is defined as the average r-TNSS score over three days of the Run-in period (2 morning (AM) and 3 evening (PM)) plus morning measurements of study day 1 (assessment in the morning prior to first administration).

SECONDARY OUTCOMES:
Mean total score change as per scale i-TNSS (AM/PM) with initial total score | Day 1, 7 and 15 post treatment
  i-TNSS (instantaneous Total Nasal Symptom Score) - TNSS scale consists of 4 symptom scores for assessment of SAR nasal symptoms (nasal congestion, rhinorrhea, nasal itching, sneezing) that reflects intensity of nasal symptoms immediately at the moment of their assessment and filling of questionnaire. Each score can be scored on a 4-point scale (0-3). Higher scores mean a more severe symptom.
  Total score as per scale i-TNSS = (Average morning score (AM) as per scale i-TNSS + Average evening score (PM) as per scale i-TNSS) / 2
  Initial total score as per scale i-TNSS = Is an average total score as per scale i-TNSS for three days of the Run-in period (2 morning (AM) and 3 evening (PM)) plus morning measurements of study day 1 (assessment in the morning prior to first administration).
Mean change in total score as per scales i-TNSS and r-TNSS with initial total score | Day 1, 7 and 15 post treatment
  Mean change in total score as per scales i-TNSS and r-TNSS with initial total score was reported.
Change in Standardized Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ(S)) | Day 1, 7 and 15 post treatment
  The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) was developed to measure the functional problems (physical, emotional, social and occupational) that are most troublesome to adults with either seasonal or perennial rhinoconjunctivitis of either allergic or non-allergic origin. RQLQ is a 7-point scale (0 = not impaired at all - 6 = severely impaired).
Number of Adverse events | throughout the study, approximately 18 days
  Number of Adverse events were reported.
Proportion of patients with at least one adverse event | throughout the study, approximately 18 days
  Proportion of patients with at least one adverse event were reported.
Proportion of patients who discontinued treatment because of an adverse event | throughout the study, approximately 18 days
  Proportion of patients who discontinued treatment because of an adverse event were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (11):
- Russia (11):
  - Sandoz Investigative Site, Chelyabinsk
  - Sandoz Investigative Site, Khasavyurt
  - Sandoz Investigative Site, Krasnodar
  - Sandoz Investigative Site, Nal'chik
  - Sandoz Investigative Site, Pyatigorsk
  - Sandoz Investigative Site, Saint Petersburg
  - Sandoz Investigative Site, Saratov
  - Sandoz Investigative Site, Stavropol
  - Sandoz Investigative Site, Vladikavkaz
  - Sandoz Investigative Site, Volgograd
  - Sandoz Investigative Site, Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.